CLINICAL TRIAL: NCT05934006
Title: Comparison of a Digital Iodine-specific Food Frequency Questionnaire With 24-hour Recall and Urinary Iodine Concentration
Brief Title: Comparison of I-FFQ and Two Reference Methods
Status: Completed | Type: Observational
Sponsor: University of Bergen (Other)
Collaborators: National Dairy Council (Other); Institute of Marine Research (Other)
Responsible Party: Sponsor
Other Study IDs: 2021/232247
Record Dates: First submitted 2023-03-06; First posted 2023-07-06 (Actual); Last update posted 2023-07-06 (Actual); Status verified 2023-07

CONDITIONS: Iodine Deficiency
Keywords: validation; food frequency questionnaire

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Biological: spot urine samples — No intervention, but measurement of urinary iodine concentration by 6 repeated spot urine samples

SUMMARY:
Mild-to-moderate iodine deficiency remains a problem in many parts of the world, including Norway. Of particular concern are fertile, pregnant, and lactating women. The Norwegian Dairy Council developed a digital iodine-specific food frequency questionnaire (I-FFQ) for the assessment of iodine intake levels, but it has yet to be validated. The main objective was thus to investigate the relative validity of the I-FFQ by comparing estimates of iodine intake obtained from the I-FFQ against a single 24-hour recall (24HR) and urinary iodine concentration (UIC) in fertile women.

ELIGIBILITY:
Inclusion Criteria:

* healthy women aged 18-40 years
* sufficient language skills to be able to complete the questionnaires in Norwegian
* be able to meet physically at the study center in Bergen

Exclusion Criteria:

* being pregnant, lactating, or having known thyroid disease

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: healthy women aged 18-40 years
Sampling Method: Non-Probability Sample
Enrollment: 72 (Actual)
Dates: Start 2021-08-10 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2022-06-15 (Actual)

PRIMARY OUTCOMES:
Comparison of FFQ with 24-hour recall | One week
  Comparison of estimated dietary iodine intake from food-frequency questionnaire (FFQ) with dietary iodine intake from 24-hour recall
Comparison of FFQ with urinary iodine concentration | One week
  Comparison of estimated iodine intake from food-frequency questionnaire (FFQ) with urinary iodine concentration (UIC)

CONTACTS AND LOCATIONS:
Overall Officials: Hanne Rosendahl-Riise, PhD, Principal Investigator — University of Bergen
Locations (1):
- University of Bergen, Bergen, Norway

IPD SHARING:
Plan to Share IPD: No